CLINICAL TRIAL: NCT02298322
Title: Study to Evaluate Non-Invasive Subcutaneous Fat Reduction in the Submental Area Using Cryolipolysis
Brief Title: Subcutaneous Fat Reduction in the Submental Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZA14-002
Record Dates: First submitted 2014-11-19; First posted 2014-11-21 (Estimated); Results first posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Body Fat Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (1):
- CoolSculpting Treatment (Experimental): The intervention is the CoolSculpting System.
  Interventions: Device: CoolSculpting System

INTERVENTIONS:
Device: CoolSculpting System

SUMMARY:
Study to Evaluate Non-Invasive Subcutaneous Fat Reduction in the Submental Area using Cryolipolysis.

Healthy adult men and women with submental skin fold thickness > 1cm who desire reduction of submental fat.

DETAILED DESCRIPTION:
Non-invasive treatment for subcutaneous fat reduction in the submental area.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects > 22 years of age and < 65 years of age.
* Submental skin fold thickness > 1cm (measured by caliper).
* No weight change exceeding 5% of body weight in the preceding month.
* Agreement to maintain his/her weight (i.e., within 5%) by not making any major changes in diet or exercise routine during the course of the study.
* Subject has signed a written informed consent form.

Exclusion Criteria:

* Skin laxity in the neck or chin area for which reduction in submental fat may, in the opinion of the investigator, result in an unacceptable aesthetic result.
* Prominent platysmal bands at rest which may interfere with assessment of submental fat
* Evidence of any cause of enlargement in the submental area other than localized subcutaneous fat, such as swollen lymph nodes or ptotic submandibular glands.
* Significant enlargement on the anterior neck that may prevent the proper placement of the applicator e.g. enlarged thyroid glands.
* Treatment with dermal fillers, radiofrequency or laser procedures, or chemical peels in the neck or chin area (below the mandible) within the past 6 months.
* Botulinum toxin or other aesthetic drug injections within the neck or chin area (below the mandible) within the past 6 months.
* History of facial nerve paresis or paralysis (such as Bell's palsy).
* History of a fat reduction procedure (e.g., liposuction, surgery, lipolytic agents, etc.) or implant in or adjacent to the area of intended treatment.
* History of prior neck surgery, or prior surgery in the area of intended treatment.
* Current dental infection.
* Known history of cryoglobulinemia, cold urticaria, or paroxysmal cold hemoglobinuria.
* Known history of Raynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
* History of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
* Currently taking or has taken diet pills or weight control supplements within the past month.
* Any dermatological conditions, such as scars in the location of the treatment area that may interfere with the treatment or evaluation.
* Active implanted device such as a pacemaker, defibrillator, or drug delivery system.
* Pregnant or intending to become pregnant in the next 6 months.
* Lactating or has been lactating in the past 6 months.
* Unable or unwilling to comply with the study requirements.
* Currently enrolled in a clinical study of an unapproved investigational drug or device.
* Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-11-11; Primary Completion 2015-08-02 (Actual); Study Completion 2015-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Brandt, BSN, Study Director — Zeltiq Aesthetics
Locations (3):
- United States (3):
  - Laser & Skin Surgery Center of Northern California, Sacramento, California
  - Zel Skin & Laser Specialists, Edina, Minnesota
  - EpiCentre Skin and Laser Center, Plano, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- CoolSculpting Treatment: Subjects treated with Coolsculpting for subcutaneous fat reduction in the submental area
Period: Overall Study
Arm/Group | CoolSculpting Treatment
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subjects treated with CoolSculpting for subcutaneous fat reduction in the submental area
Groups:
- CoolSculpting Treatment: Subjects treated with CoolSculpting for fat reduction in the submittal area
Arm/Group | CoolSculpting Treatment
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 49.3 [25 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Safety of CoolScupting in the Submental Area
Description: Safety of the Zeltiq CoolSculpting device will be assessed by measuring the incidence of device- and/or procedure-related adverse events. Adverse event reports are collected from the time of enrollment through the 12 week follow-up visit.
Time Frame: Time of enrollment through12 week post-final treatment follow-up
Population: As-treated population of 60 subjects who received CoolSculpting treatment for subcutaneous fat reduction in the submental area.
Measure: Number; unit: incidence of device- and/or procedure AE
Arm/Group | CoolSculpting Treatment
Number analyzed (Participants) | 60
incidence of device- and/or procedure AE | 4

2. Primary Outcome: Percentage of Correct Identification of Pre-treatment Photographs
Description: Change in the treated vs. untreated areas will be assessed by observation of changes in surface contour and/or fat volume by an independent photo review of pre-treatment and post-treatment images of the treated areas. Reviewers will be practicing dermatologists or plastic surgeons. All reviewers will be blinded to post-treatment vs. baseline untreated area. The order in which images will be presented will be randomized; for each subject placement of the baseline, pre-treatment image will be randomized for each pair of subject images. Reviewers will be asked to select the baseline photos for each subject photo series and record selections on a data collection form. Criteria for evaluable photos for the purposes of the independent review: subject completed treatment regimen; subject has complete set of baseline photos; subject has a complete set of post-treatment photos; photos were taken using Zeltiq standard procedure.
Time Frame: 12 week post-final-treatment
Population: Subjects included in the analysis group (58) received full treatment; treatment was interrupted for 2 subjects not included in this population.
Measure: Number; unit: percentage of correcty identified photos
Units Other Than Participants: photo pairs
Groups:
- CoolSculpting Treatment: Per-protocol subjects treated with CoolSculpting for fat reduction in the submental area
Arm/Group | CoolSculpting Treatment
Number analyzed (Participants) | 58
Number analyzed (photo pairs) | 58
percentage of correcty identified photos | 91.4
Statistical Analysis 1: Comparison: CoolSculpting Treatment; Test type: Other; p < 0.0001, t-test, 1 sided; sucess proportion = 91.4, 95% CI 2-sided [86.2 to 95.1]

3. Secondary Outcome: Change in the Fat Layer of the Treated Area as Measured by Ultrasound
Description: Change in the fat layer thickness will be calculated by comparison of pre-treatment and 16 week post-treatment ultrasound measurements taken in the area treated with the device. The Sponsor's standardized techniques for obtaining ultrasound imaging will be used. Results indicate the fat layer reduction in cm.
Time Frame: 12 weeks post-final treatment
Population: Evaluable ultrasound images were available for 57 of the 59 subjects completing the 12 week follow-up visit.
Measure: Mean (Standard Deviation); unit: cm fat layer reduction post-procedure
Groups:
- CoolSculpting Treatment: Subjects with CoolSculpting treatment for subcutaneous fat reduction of the submental area
Arm/Group | CoolSculpting Treatment
Number analyzed (Participants) | 57
cm fat layer reduction post-procedure | -0.20 (0.19)

4. Secondary Outcome: Subject Satisfaction With CoolScupting in the Submental Area
Description: Subject satisfaction as assessed by questionnaires administered at 12 weeks post-final treatment. The questionnaire will ask the subject about their treatment experience and the efficacy of the treatment.
Time Frame: 12 weeks post-final treatment
Population: As-treated population of subjects who received CoolSculpting for subcutaneous fat reduction of the submental area who completed a Subject Satisfaction Questionnaire at the 12-week final follow-up visit.
Measure: Count of Participants; unit: Participants
Groups:
- CoolSculpting Treatment: As-treated population of subjects who received CoolSculpting for subcutaneous fat reduction of the submental area who completed a Subject Satisfaction Questionnaire at the 12-week final follow-up visit.
Arm/Group | CoolSculpting Treatment
Number analyzed (Participants) | 60
Participants
  Visible/Very Visible Fat Reduction | 46
  Satisfied/VerySatisfied with CoolSculpting | 50
  Procedure was Very Comfortable/Comfortable | 45
  Strongly Agree/Agree Procedure made more youthful | 30
  Strongly Agree/Agree chin looked more toned | 45
  Strongly Agree/Agree appearance has improved | 46
  Effect from procedure More Than Expected/Expected | 40
  Would recommend procedure to a friend | 48
  Feel less self-conscious about chin fat | 43

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from enrollment through the 12-week final follow-up visit.
Description: Anticipated deaths = 0 participants Unanticipated deaths = 0 participants
Arm/Group | CoolSculpting Treatment
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 2/60
Other Adverse Events (participants affected / at risk) | 15/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CoolSculpting Treatment (N=60)
Food poisoning (Gastrointestinal disorders) | 1 (1) — Food poisoning reported as moderate in severity. No relationship to CoolSculpting System or procedure.
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Skin cancer on back, reported as severe. Not related to CoolSculpting System or procedure.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CoolSculpting Treatment (N=60)
Pinched nerve (Musculoskeletal and connective tissue disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Broken finger (Musculoskeletal and connective tissue disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Torn meniscus (Musculoskeletal and connective tissue disorders) | 1 (1)
Hives (General disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Cold (General disorders) | 5 (5)
Prolonged erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Cold sore (General disorders) | 1 (1)
Hyper pigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Breast infection (Infections and infestations) | 1 (1)
Back of throat fullness sensation (General disorders) | 1 (1)
Food Poisoning (Gastrointestinal disorders) | 1 (1)
Skin cancer (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No